CLINICAL TRIAL: NCT07252505
Title: Early Intravenous Magnesium Sulfate and Its Impact on Cerebral Vasospasm in Traumatic Subarachnoid Hemorrhage
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Salah El-Dein Quashty Aly, Emergency Medicine assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Magnesium Sulfate
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Trauma and Emergency Care
MeSH Terms: conditions — Wounds and Injuries | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: patients will be given magnesium sulfate (MgSO4) with infusion rate (20- 40 mmol) per hour. (Placebo Comparator): will be given magnesium sulfate (MgSO4) with infusion rate (20- 40 mmol)
  Interventions: Drug: Magnesium Sulfate 10 MG/ML
- Group B: will be given normal saline (placebo group). (No Intervention): will be given normal saline (placebo group).

INTERVENTIONS:
Drug: Magnesium Sulfate 10 MG/ML — As a rule, MgSO4 will be given(for group A) within 24 hours after establishing a diagnosis of tSAH. The protocol will include MgSO4 10% application with a loading dose of 50 mg/kg body weight over 1 hour. The infusion rate (20-40 mmol) per hour will depend on blood pressure with a target mean arterial pressure of 65 mm Hg. Thereafter, patients will receive a continuous application of 81 mmol/ 24 hours for a maximum of 7 days. Target Serum Magnesium Levels Serum magnesium levels will be monitored daily during the infusion period. The target therapeutic range for serum magnesium will be between 2.0-2.5 mmol/L. If the serum magnesium level exceeds the upper limit (2.5 mmol/L), the infusion rate will be reduced, and the patient will be closely monitored for signs of magnesium toxicity, such as hypotension, bradycardia, respiratory depression, or reflexes loss. In the event of severe hyper-magnesemia, calcium gluconate will be administered as an antidote.
  Other Names: MgSo4
  Arms: Group A: patients will be given magnesium sulfate (MgSO4) with infusion rate (20- 40 mmol) per hour.

SUMMARY:
Subarachnoid hemorrhage (SAH) is a clinical phenomenon caused by the abrupt rupture and bleeding of blood vessels at the surface or base of the brain, which can occur for a number of reasons. As a result, the subarachnoid membrane receives direct blood flow. SAH is a debilitating neurological disorder with high morbidity and mortality. Despite advancements in medicine and surgical care, patients who survive their first bleeding event are at high risk for secondary sequelae, including delayed cerebral ischemia (DCI) and cerebral vasospasm (CV)

CV denotes a temporary, self-resolving constriction of the intracranial arteries that occurs several days after an SAH. This phenomenon is closely linked to clinical deterioration resulting from DCI, affecting up to 30% to 40% of patients. DCI is a significant clinical event that typically manifests 3 to 14 days after the initial bleeding and is characterized by subsequent neurological deterioration. These complications can lead to poor functional outcomes and long-term disability

Subarachnoid hemorrhage is classified into aneurysmal subarachnoid hemorrhage (aSAH) and Traumatic SAH (tSAH). TSAH has been described as an adverse prognostic factor leading to progressive neurological deterioration and increased morbidity and mortality. Traumatic subarachnoid hemorrhage is caused by head injuries from events like falls, motor vehicle crashes, and blows to the head, which damage blood vessels within the skull. The injury itself is the primary cause, leading to the brain being hit against the skull and tearing these blood vessels

DETAILED DESCRIPTION:
Magnesium is a noncompetitive calcium antagonist with several important vascular and potentially neuro-protective effects. For instance, magnesium can lead to vasodilatation by blocking the voltage-dependent calcium channel and decreasing glutamate release and block the influx of calcium ions, inhibiting blood vessel contraction and preventing CV.In addition, magnesium also attenuates the effect of various potent vasoconstrictors, such as endothelin 1, and blocks the formation of reactive oxygen species These potentially helpful effects of magnesium on vasodilation and consequent neuro-protection has led some investigators to study the ability of magnesium to prevent of cerebral vasospasm and delayed cerebral ischemia after subarachnoid hemorrhage (SAH). Limited data exist for tSAH. Early intravenous Magnesium Sulfate (MgSO₄)application within 24 hours after diagnosis may prevent or attenuate vasospasm and improve neurological recovery and outcome

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between eighteen to sixty five years Diagnosed with tSAH on Head Computed Tomography(CT)within 24 hours of trauma.
* Both Genders are included Indication for endovascular or microsurgical treatment plan

Exclusion Criteria:

* Aneurysmal or spontaneous SAH Sever hepatic dysfunction.
* Known hypersensitivity to magnesium sulfate
* Renal disease with glomerular filtration rate<15 ml/min.
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of early intravenous magnesium sulfate on the incidence and severity of cerebral vasospasm in patients with traumatic subarachnoid hemorrhage assessed by cerebral blood flow velocity measured Through Transcranial Doppler | From Day 1 immediately poat trauma (baseline) till an average of 7 Days".
  To evaluate the effect of early intravenous magnesium sulfate on the incidence and severity of cerebral vasospasm in patients with traumatic subarachnoid hemorrhage assessed by cerebral blood flow velocity measured Through Transcranial Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Quashty, MD, Principal Investigator — Assisstant lecturer

IPD SHARING:
Plan to Share IPD: No